CLINICAL TRIAL: NCT05556239
Title: The Effect of Resistance Training in Patients With Malignant Lymphoma Undergoing Chemotherapy Treatment - the STAY STRONG TRIAL - a Randomized Controlled Trial.
Brief Title: STAY-STRONG Study of Exercise Training During Chemotherapy
Acronym: STAY-STRONG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jan Christensen, Senior researcher, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-22014826
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma, B-Cell; Lymphoma, Hodgkin; Exercise; Body Composition; Physical Functional Performance; Quality of Life; Sarcopenia; Muscle, Skeletal; Patient Reported Outcome Measures
MeSH Terms: conditions — Lymphoma, B-Cell; Hodgkin Disease; Motor Activity; Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The usual care group (No Intervention): The usual care group receives standard care in accordance to current clinical practice at Rigshospitalet
- Resistance Exercise Training (Experimental): Patients included in the intervention group will receive usual care plus the exercise training intervention.
  Interventions: Behavioral: Resistance Exercise Training

INTERVENTIONS:
Behavioral: Resistance Exercise Training — Supervised resistance training program planned as 3 sessions per week of approximately 60 minutes. The resistance training program comprises 6 exercises for the major muscle groups, starting at 2 sets of 15 repetitions maximum progressing to 4 sets of 8 repetitions maximum. Each session will be supervised by physiotherapist to ensure proper technique, and progression in training load. The participants will choose an exercise ambassador from their network, who during the period will be encouraged to, on a weekly basis, to be in contact with the participant.
  Arms: Resistance Exercise Training

SUMMARY:
This study evaluates the effectiveness of a supervised progressive resistance training program in patients malignant lymphomas with the primary outcome being lean body mass.

The study is designed as a a single center, two-armed, parallel-group, investigator-initiated clinical randomized controlled superiority trail evaluating the effectiveness of a 4-month supervised progressive resistance training intervention compared to usual care.

DETAILED DESCRIPTION:
New approaches of early rehabilitation are needed to maintain physical function levels in patients with malignant lymphoma patients during chemotherapy treatment. The STAY STRONG TRAIL has the potential to become the future model of care and rehabilitation with the prospect of reducing the complex symptom burden, supporting treatment tolerance, maintaining physical function and, by extension, improve the patient's chances of survival and quality of life. This study will be among the first to include structured and supervised progressive resistance training during the complete 1st line anthracycline-containing combination chemotherapy regime in patients treated with Diffuse Large B-Cell Lymphoma and Hodgkin Lymphoma.

At present, there is a lack of knowledge regarding the potential effect of exercise to counteract muscle atrophy during chemotherapy in patients with malignant lymphomas. The overall aim of the present STAY STRONG TRAIL is to investigate whether a structured and supervised progressive resistance training program during the complete first line anthracycline-containing combination chemotherapy with support from an 'exercise ambassador' can preserve muscle function and prevent muscle dysfunction in patients newly diagnosed with Diffuse Large B-Cell Lymphoma and Hodgkin Lymphoma referred to first line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must:

  * Be newly diagnosed with diffuse large B-cell lymphoma and Hodgkin Lymphoma
  * Be expected to receive treatment with an anthracycline-containing combination chemotherapy at the Department of Hematology, Rigshospitalet
  * Be ≥ 18 years of age at the time of signing the informed consent form.
  * Be residing in Denmark
  * Have an Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2
  * Be able to speak and read Danish, and to provide a signed informed consent form.

Exclusion Criteria:

* Patients with:

  * Clinically significant cardiovascular disease, including, but not limited to: Heart failure NYHA (New York Heart Association) class III-IV, uncontrolled hypertension, and symptomatic cardiac arrhythmias.
  * Psychiatric, neurological, or geographical conditions that could influence protocol adherence.
  * Disorders that cause an inability to perform exercise training for one hour.
  * Any other known malignancy requiring active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Lean Body Mass | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Change in lean body mass. Assessed by whole-body dual-energy x-ray absorptiometry (DXA) scan.

SECONDARY OUTCOMES:
Functional performance: Habitual gait speed | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in habitual gait speed. Assessed using a 10-Meter walk test
Functional performance: Maximal gait speed | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in maximal gait speed assessed using a 10-Meter walk test
Functional performance: Stair climbing power | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in stair climbing power following a fixed protocol.
Functional performance: Sit-to-stand | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in Sit-to-stand performance is evaluated by the 30-seconds Sit-to-Stand Test (30s STS)
Muscle strength:Hand grip strength | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in Hand grip strength. Assessed by a dynamometer
Muscle strength:Maximal isometric knee extensor strength | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in maximal isometric knee extensor strength. Assessed by a dynamometer
Leg-extensor power | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in maximum leg power assessed by Nottingham Power Rig
Health Related Quality of Life | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in patient-reported health-related quality of life assessed using the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire EORTC (EORTC-QLQ-C30)
Symptoms burden | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in patient-reported symptoms burden assessed using the in M.D. Anderson Symptom Inventory questionnaire (MDASI)
Depression and Anxiety. | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in patient-reported depression and anxiety, assessed using the Hospital Anxiety and Depression Scale (HADS).
Leisure time physical activity | Baseline, 4-month follow-up
  Changes in leisure time physical activity. Assessed by activity accelerometer (ActiGraph wGT3x-BT). Participants will be instructed to wear the accelerometer at their waist for 24 h during ten consecutive days.
Inflammation marker: Tumor necrosis factor alpha (TNF- α) | Baseline, 4-month follow-up
  Changes in blood TNF- α concentration
Inflammation marker: interleukin (IL)-13 | Baseline, 4-month follow-up
  Changes in blood IL-13 concentration
Inflammation marker: Interleukin (IL)-6 | Baseline, 4-month follow-up
  Changes in blood IL-6 concentration
Inflammation markers: High-sensitivity C-reactive Protein (hsCRP) | Baseline, 4-month follow-up
  Changes in blood hsCRP concentration
Biomarker of muscle atrophy and muscle wasting: Growth differentiation factor 11 (GDF11) | Baseline, 4-month follow-up
  Changes in blood GDF11 concentration
Biomarker of muscle atrophy and muscle wasting: Growth differentiation factor 15 (GDF15) | Baseline, 4-month follow-up
  Changes in blood GDF15 concentration
Body composition and anthropometrics: Fat percentage | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in whole-body fat percentage assessed by DXA scan.
Body composition and anthropometrics: Body mass | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in body mass
Body composition and anthropometrics: Total fat mass | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in total fat mass, assessed by DXA
Body composition and anthropometrics: Body mass index (BMI) | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in BMI. Weight will be measured by scale (kg). Height will be measured by measuring (m). BMI will be derived from weight and height (kg/m^2)
Exercise feasibility: Exercise sessions attendance rate | From baseline to 4-month follow-up
  Exercise sessions attendance rate (%), defined as number of attended exercise sessions / number of prescribed exercise sessions x 100
Exercise feasibility: Patient-reported symptomatic adverse events (pain, dizziness, nausea, fatigue, other) | Immediately before and immediately after each exercise session performed from baseline to 4-month follow-up
  Changes in patient-reported symptomatic adverse events (pain, dizziness, nausea, fatigue, other)

OTHER OUTCOMES:
Muscle biopsies | Baseline, 4-month follow-up
  Muscle biopsies will be taken on a selected number of subjects from the vastus lateralis muscle, for the use in future analysis of i.e. muscle fibre size and distribution, myogenic stem cell activity,
Muscle Architecture: Muscle Thickness | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in muscle thickness will be assessed by ultrasound imaging.
Muscle Architecture: Pennation Angle | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in pennation angle will be assessed by ultrasound imaging.
Self-reported physical activity | Baseline
  Changes in patient-reported weekly duration of physical activity assessed using The International Physical Activity Questionnaires (I-PAQ, short form)
Nutrition | Baseline, 4-month follow-up, 8-month follow-up, 1-year follow-up
  Changes in patient-reported nutritional status assessed using The Short Nutritional Assessment Questionnaire (SNAQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939